CLINICAL TRIAL: NCT02381912
Title: Sexual Function in Patients Suspected of Non-muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Peter Busch Østergren, MD, Herlev Hospital
Other Study IDs: SSBC-2015
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Bladder Neoplasms; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Erectile Dysfunction; Hematuria
MeSH Terms: conditions — Urinary Bladder Neoplasms; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Erectile Dysfunction; Hematuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hematuria - NMIBC: Primary hematuria due to NMIBC.
  Interventions: Other: EORTC QLQ-C30 and EORTC BLS-24 questionnaire
- Hematuria - other cause: Other non-malignant cause of hematuria.
  Interventions: Other: EORTC QLQ-C30 and EORTC BLS-24 questionnaire

INTERVENTIONS:
Other: EORTC QLQ-C30 and EORTC BLS-24 questionnaire — Questionnaires answered at baseline and 4 months follow up.

SUMMARY:
The purpose of the study is to investigate sexual function in patients suspected of non muscle invasive bladder cancer (NMIBC). The investigators hypothesis is that reduced sexual function is underdiagnosed in patients with non-muscle invasive bladder cancer and that active examination and treatment may worsen the sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hematuria, both gross and microscopic
* Men and women older or equal to 40 years of age
* Signed informed consent statement

Exclusion Criteria:

* Men and women younger than 40 years of age
* Patients with recurrent hematuria and known causative disease
* Already known urogenital cancer
* Previous massive pelvic surgery or pelvic radiotherapy
* TUR-P within the last 2 months
* Participants diagnosed with tumors originating from the ureters, renal pelvis and kidney, and bladder tumors at T stage more than or equal to T1b.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hematuria.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in sexual function | 4 months
  Change in sexual function measured by the "EORTC QLQ-BLS24 sexual functioning questions"

SECONDARY OUTCOMES:
Change in erectile function | 4 months
  Change in erectile function measured by the Erection Hardness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Østergren, MD, Principal Investigator — Herlev Hospital, Department of Urology
Locations (1):
- Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Background] Kowalkowski MA, Chandrashekar A, Amiel GE, Lerner SP, Wittmann DA, Latini DM, Goltz HH. Examining sexual dysfunction in non-muscle-invasive bladder cancer: results of cross-sectional mixed-methods research. Sex Med. 2014 Aug;2(3):141-51. doi: 10.1002/sm2.24. PMID 25356311
- [Background] van der Aa MN, Bekker MD, van der Kwast TH, Essink-Bot ML, Steyerberg EW, Zwarthoff EC, Sen FE, Elzevier HW. Sexual function of patients under surveillance for bladder cancer. BJU Int. 2009 Jul;104(1):35-40. doi: 10.1111/j.1464-410X.2008.08333.x. Epub 2009 Jan 14. PMID 19154473
- [Background] Goossens-Laan CA, Kil PJ, Ruud Bosch JL, De Vries J. Pre-diagnosis quality of life (QoL) in patients with hematuria: comparison of bladder cancer with other causes. Qual Life Res. 2013 Mar;22(2):309-15. doi: 10.1007/s11136-012-0163-1. Epub 2012 Mar 30. PMID 22461137